CLINICAL TRIAL: NCT04084652
Title: Comparing the Muscle Protein Synthetic Response to Ingestion of Mycoprotein vs Protein Isolated From Mycoprotein
Brief Title: Mycoprotein and Muscle Protein Synthetic Response
Acronym: PIMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Quorn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 190206/B/07UOE
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Anabolic Response to Mycoprotein and Micronutrient Ingeston

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mycoprotein (Experimental): Mycoprotein in its full food matrix
  Interventions: Dietary Supplement: Mycoprotein ingestion
- Protein Isolated from Mycoprotein (Experimental): Protein from mycoprotein isolated from the food matrix
  Interventions: Dietary Supplement: Mycoprotein ingestion

INTERVENTIONS:
Dietary Supplement: Mycoprotein ingestion — The ingestion of mycoprotein

SUMMARY:
Dietary protein is vital for the preservation of health and optimal adaptation to training. However, traditional animal proteins come with a number of economic, environmental, and ethical issues. Accordingly, there is a need to develop an understanding of the utility of more sustainable non-animal derived dietary proteins to support our nutrition. Mycoprotein, produced by Quorn Foods™, has recently been shown to stimulate a greater anabolic response within skeletal muscle compared with milk protein, suggesting its utility within sports nutrition. However, it is unclear what accounted for the greater anabolic response of mycoprotein. One explanation could be the non-protein nutrients contained within mycoprotein (e.g. fibre, carbohydrate, fat or micronutrients).

Therefore, the present study will compare the muscle anabolic response between mycoprotein (MYC) as a whole food and the protein isolated from mycoprotein (PIM).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30.
* Resistance trained

Exclusion Criteria:

* Any metabolic impairments.
* Cardio/pulmonary diseases.
* Chronic use of over the counter pharmaceuticals
* A personal or family history of epilepsy, seizures or schizophrenia.
* Allergic to mycoprotein/Quorn/edible fungi/environmental mould products.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 7.5 hours
  The rate of synthesis of new muscle protein (Fractional Synthetic Rate %/h)

SECONDARY OUTCOMES:
Plasma Amino Acid Kinetics | 7.5 hours
  The rate of appearance of amino acids ingested in the drink
Blood Glucose | 7.5 hours
  The levels of glucose in the blood
Serum Insulin | 7.5 hours
  The levels of insulin in blood serum

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No